CLINICAL TRIAL: NCT05696717
Title: A Phase 3, Multi-center, Randomized Withdrawal and Long Term Extension Study of Ampreloxetine for the Treatment of Symptomatic Neurogenic Orthostatic Hypotension in Participants With Multiple System Atrophy
Brief Title: Phase 3 Efficacy and Durability of Ampreloxetine for the Treatment of Symptomatic nOH in Participants With Multiple System Atrophy
Acronym: CYPRESS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-003903-14
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-11

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension; MSA - Multiple System Atrophy
MeSH Terms: conditions — Shy-Drager Syndrome | interventions — ampreloxetine

STUDY DESIGN:
Intervention Model Description: Open Label followed by Randomized Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ampreloxetine (Open Label) (Active Comparator): Participants will receive ampreloxetine as a single, oral, daily dose of active drug for 12 weeks.
  Interventions: Drug: Ampreloxetine
- Ampreloxetine (Randomized Withdrawal) (Placebo Comparator): After completing the open label, participants are randomized to either ampreloxetine or placebo receiving a single, oral, daily dose of active drug or placebo for a further 8 weeks.
  Interventions: Drug: Ampreloxetine; Drug: Placebo
- Long-Term Extension Period (Active Comparator): Participants will receive ampreloxetine as a single, oral, daily dose of active drug for 104 weeks.
  Interventions: Drug: Ampreloxetine

INTERVENTIONS:
Drug: Ampreloxetine — Oral tablet, QD
  Other Names: TD-9855
Drug: Placebo — Oral tablet, QD
  Arms: Ampreloxetine (Randomized Withdrawal)

SUMMARY:
This is a Phase 3, multi-center, randomized withdrawal study to evaluate the efficacy and durability of ampreloxetine in participants with MSA and symptomatic nOH after 20 weeks of treatment. This study includes 4 periods: Screening, open label, randomized withdrawal, and long-term treatment extension (LTE).

ELIGIBILITY:
Inclusion Criteria:

* Participant is male or female and at least 30 years old.
* Participant has a diagnosis of possible or probable MSA of the Parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) according to The Gilman Criteria (2008).
* Participant has a diagnosis of possible or probable MSA of the Parkinsonian subtype (MSA-P) or cerebellar subtype (MSA-C) confirmed by the Enrollment Steering Committee (ESC).
* Participant must meet the diagnostic criteria of nOH, as demonstrated by a sustained reduction in BP of ≥20 mmHg (systolic) or ≥10 mmHg (diastolic) within 3 min of standing as part of orthostatic standing test or being tilted up ≥60o from a supine position as determined by a tilt-table test.
* Participant must score ≤4 on UMSARS Part IV at Visit 1 (Screening).
* Participant must score at least a 4 on the OHSA item 1 at Visit 2 (Day 1).
* Participant must be willing to not take any prohibited medications during the study.
* If participant is female, the participant must not be pregnant, breastfeeding, or planning a pregnancy during the course of the study. A woman of childbearing potential must have a documented negative pregnancy test at screening.
* During the study and for 30 days after receiving the last dose of the study drug, females of childbearing potential or males capable of fathering children must agree to use highly effective birth control measures (failure rate <1% when used consistently and correctly) or agree to abstain from sexual intercourse.
* Participant is willing and able to provide signed and dated written informed consent to -participate prior to initiation of any study related procedures.

Participant is able to communicate well with the Investigator and clinic staff, understands the expectations of the study and is able to comply with the study procedures, requirements, and restrictions.

Exclusion Criteria:

* Participant has a systemic illness known to produce autonomic neuropathy, including, but not limited to, amyloidosis and autoimmune neuropathies. Participant with diabetes mellitus (DM) will be evaluated on a case-by-case basis by the medical monitor and considered ineligible unless they meet all of the following criteria:

  * Well controlled type-2 DM in treatment with only oral medications and diet
  * HbA1C of ≤7.5% performed during screening or up to 12 weeks before screening
  * No clinically evident peripheral neuropathy (e.g., normal sensory examination on peripheral extremities)
  * No known retinopathy (e.g., annual ophthalmic exam is sufficient)
  * No nephropathy (e.g., absence of albuminuria and GFR >60).
* Participant has a known intolerance to other NRIs or SNRIs.
* Participant currently uses concomitant antihypertensive medication for the treatment of essential hypertension.
* Participant has used strong CYP1A2 inhibitors or inducers within 7 days or 5 half lives, whichever is longer, prior to Visit 2 (Day 1) or requires concomitant use until the Safety follow-up Visit.
* Participant has changed dose, frequency, or type of prescribed medication for orthostatic hypotension within 7 days prior to Visit 2 (Day 1).
* Midodrine and droxidopa (if applicable) must be tapered off and stopped at least 7 days prior to Visit 2 (Day 1).
* Participant has known or suspected alcohol or substance abuse within the past 12 months (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision [DSM IV TR®] definition of alcohol or substance abuse).
* Participant has clinically unstable coronary artery disease or had a major cardiovascular event (e.g., myocardial infarction) in the past 6 months.
* Participant has significant uncontrolled cardiac arrhythmia, history of complete heart block, or significant QTc prolongation (≥450 msec for males and ≥470 msec for females).
* Participant has a new onset of a neurological event (i.e., seizures, confusion, altered levels of consciousness, etc.) in the past 6 months.
* Participant has used any monoamine oxidase inhibitor (MAOI) within 14 days prior to Visit 2 (Day 1).
* Participant has a history of untreated closed angle glaucoma, or treated closed angle glaucoma that, in the opinion of an ophthalmologist, might result in an increased risk to the participant.
* Participant has a Montreal Cognitive Assessment (MoCA) <21.
* Participant is unable or unwilling to complete all protocol specified procedures including questionnaires.
* Participant has known congestive heart failure (New York Heart Association [NYHA] Class 3 or 4).
* Participant has had any malignant disease, other than carcinoma in situ of the cervix or basal cell carcinoma, within the past 2 years prior to Screening.
* Participant has a known gastrointestinal (GI) condition, which in the Investigator's judgment, may affect the absorption of study medication (e.g., ulcerative colitis, gastric bypass).
* Participant has psychiatric, neurological, or behavioral disorders that may interfere with the cognitive ability of the participant to give informed consent, understand and comply with study procedures, or interfere with the conduct of the study.
* Participant is currently receiving any investigational drug or has received an investigational drug within 30 days of dosing. An investigational drug is defined as a drug that is not approved by a regulatory agency (e.g., Food and Drug Administration [FDA]).
* Participant has a clinically significant abnormal laboratory finding(s) (e.g., alanine aminotransferase [ALT] or aspartate aminotransferase [AST] ≥3.0 x upper limit of normal [ULN]; blood bilirubin [total] ≥3.0 x ULN; estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or any abnormal laboratory value that could interfere with safety of the participant).
* Participant has demonstrated lifetime suicidal ideation and/or suicidal behavior, as outlined by the C-SSRS (Baseline/Screening Version). Participant should be assessed by the rater for risk of suicide and the participant's appropriateness for inclusion in the study.
* Participant has a concurrent disease or condition (e.g., COVID-19), or recent surgery, that in the opinion of the Investigator, would confound or interfere with study participation or evaluation of safety, tolerability, or absorption of the study drug.
* Participant has known hypersensitivity to ampreloxetine (ampreloxetine hydrochloride), or any excipients in the formulation.
* Major surgery (i.e., procedures involving higher risk for infection and extended recovery period, such as, joint replacement, gastric bypass, open heart surgery, organ transplant, etc.) occurring less than 4 weeks prior to enrollment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in OHSA composite score at Week 8 during the double-blind RW period | 8-week randomized withdrawal period (Week 12 to Week 20)
  Score change from baseline on the composite of Questions 1 - 6 of the Orthostatic Hypotension Symptom Assessment (OHSA).

SECONDARY OUTCOMES:
Change from baseline in OHDAS item 1 (activities that require standing for a short time) at Week 8 post randomization | 8-week randomized withdrawal period (Week 12 to Week 20)
  Orthostatic Hypotension Daily Activities Scale (OHDAS) is an assessment of how low blood pressure symptoms affect daily life.
Change from baseline in OHDAS item 3 (activities that require walking for a short time) at Week 8 post randomization | 8-week randomized withdrawal period (Week 12 to Week 20)
  Orthostatic Hypotension Daily Activities Scale (OHDAS) is an assessment of how low blood pressure symptoms affect daily life.

CONTACTS AND LOCATIONS:
Locations (79):
- United States (26):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - UC San Diego Movement Disorder Center, La Jolla, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinson's Disease And Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - SFM Clinical Research, LLC, Boca Raton, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Neurostudies, Inc, Port Charlotte, Florida
  - University of South Florida Ataxia Research Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Health System, Glenview, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Brigham and Women's Hospital (Neuromuscular Division), Boston, Massachusetts
  - Massachusetts Chan Medical School, Worcester, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - NYU Langone Health NYU Dysautonomia Center, New York, New York
  - The Neurological Institute at Columbia University Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Movement Disorders and Autonomic Disorders Clinic; University of Utah, Salt Lake City, Utah
- Argentina (6):
  - INEBA Instituto Neurociencias Buenos Aires, CABA, Buenos Aires F.D.
  - Instituto Fleni, CABA, Buenos Aires F.D.
  - Médico/Hospital de la Policía Federal Churruca Visca, CABA, Buenos Aires F.D.
  - Hospital General de Agudos Jose Maria Ramos Mejía, CABA
  - Hospital Británico de Buenos Aires, CABA
  - Fundación Scherbovsky, Mendoza
- Australia (3):
  - Monash Health, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Theravance Biopharma Investigative Site, Parkville, Victoria
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Universitatsklinikum Tulln, Tulln
- Brazil (4):
  - Instituto de Neurologia de Curitiba S\C LTDA, Curitiba, Paraná
  - Hospital de Clínicas - Universidade Federal de Minas Gerais (HC - UFMG), Belo Horizonte
  - Centro de Pesquisa Clínica (CPC) do Hospital das Clínicas de Porto Alegre (HCPA), Porto Alegre
  - Hospital São Lucas - PUCRS, Porto Alegre
- University of Calgary - Health Sciences Centre, Calgary, Alberta, Canada
- Bispebjerg Hospital, Copenhagen, Denmark
- Estonia (2):
  - Astra Clinic (Clinic4U), Tallinn
  - Tartu University Hospital, Tartu
- France (3):
  - Hopital Caremeau, Nîmes, Occitanie
  - Centre Hospitalier Universitaire de Bordeaux Health, Bordeaux
  - Centre d'Investigation Clinique Hôpital Pierre Paul Rique, Toulouse
- Germany (3):
  - Praxis Dr. Oehlwein, Outpatient Clinic, Gera, Thuringia
  - Charité - Universitätsmedizin Berlin- Campus Mitte, Berlin
  - Charite Universitaetsmedizin Berlin, Berlin
- Semmelweis Egyetem, Budapest, Hungary
- Theravance Biopharma Investigative Site, Tel Aviv, Israel
- Italy (8):
  - IRCCS Istituto de Scienze Neurologiche di Bologna (ISNB), Bologna
  - Parkinson's Centre of Ospedale CTO, Milan
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno, Salerno
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Santa Chiara Hospital, Trento
  - Pia Fond. Cardinale Giovanni Panico Azienda Ospedaliera, Tricase
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Theravance Biopharma Investigative Site, Christchurch
- Poland (4):
  - Neurocentrum-Miwomed, Gdansk
  - Neuro-Care Sp. z o.o. Sp. Komandytowa, Katowice
  - Krakowska Akademia Neurologii Sp.zo.o., Krakow
  - Instytut Zdrowia dr Boczarska-Jedynak Sp. z o.o., Sp.k., Oświęcim
- CNS-Campus Neurologico Senior, Torres Vedras, Portugal
- University of Belgrade Neurology Clinic, Belgrade, Serbia
- Spain (5):
  - Fundació Assistencial Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Germans Trias i Pujol, Department of Neurology, Barakaldo, Bizkaia
  - Instituto Investigación Sanitaria Biocruces, Barakaldo, Bizkaia
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Infante Sofia Paseo Europa, Madrid
- National Taiwan University Cancer Center, Taipei, Taiwan, Taiwan
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health, London
  - Autonomic Unit, National Hospital for Neurology & Neurosurgery, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: No